CLINICAL TRIAL: NCT07038902
Title: A Comparative Study Between Modified Miniscrew-Assisted Rapid Palatal Expander And Modified Rapid Palatal Expander in Molar Distalization Using Cone- Beam Computed Tomography
Acronym: MIDPAC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Marwa Abd ELhamid Ahmed Abu Elhagag, Principal Investigator, Clinical Researcher, Al-Azhar University (Assiut branch), Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMARPE-MRPE-CBCT-DISTAL2025-AZ; MIDPAC-AZU-2025 (Registry Identifier: Clinical Trials.gov)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Malocclusion, Class I/II; Crowding; Maxillary First Molar Distalization
Keywords: Modified MARPE; Modified RPE; Molar Distalization; CBCT; Orthodontics
MeSH Terms: conditions — Malocclusion; Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Miniscrew-Assisted Rapid Palatal Expander (MARPE) (Experimental)
  Interventions: Device: Group A: Modified Miniscrew-Assisted Rapid Palatal Expander (MARPE)
- Modified Rapid Palatal Expander (RPE) (Experimental)
  Interventions: Device: Group B: Modified Rapid Palatal Expander (RPE)

INTERVENTIONS:
Device: Group A: Modified Miniscrew-Assisted Rapid Palatal Expander (MARPE) — A skeletal anchorage-supported with miniscrews inserted into the palate using a self-drilling technique.
  Arms: Modified Miniscrew-Assisted Rapid Palatal Expander (MARPE)
Device: Group B: Modified Rapid Palatal Expander (RPE) — A tooth-borne anchorage focusing on molar distalization .
  Arms: Modified Rapid Palatal Expander (RPE)

SUMMARY:
Comparative study between modified miniscrew-assisted rapid palatal expander and modified rapid palatal expander in molar distalization using CBCT.

DETAILED DESCRIPTION:
This research will be conducted as a prospective and randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Presence of permanent dentition
* Skeletal Class I
* Dental Class II molar relationship with moderate dental crowding
* Crowding >4mm
* Good oral hygiene
* Healthy periodontal condition

Exclusion Criteria:

* Presence of craniofacial syndromes or cleft palate
* History of previous orthodontic treatment
* Poor oral hygiene or active periodontal disease
* Contraindications to CBCT imaging (e.g., pregnancy, inability to remain still during the scan)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Amount of Molar Distalization Measured by CBCT | Baseline (prior to initiation of molar distalization) At the end of the molar distalization phase (approximately 12 weeks post-treatment initiation).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Ahmed Salim, Professor, Study Director — Department of Orthodontics, Faculty of Dental Medicine, Al-Azhar University, Assiut branch.
Locations (1):
- Department of Orthodontics, Faculty of Dental Medicine, Al-Azhar University, Assiut branch., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided